CLINICAL TRIAL: NCT00583050
Title: Endovascular Exclusion of Thoracoabdominal Aortic Aneurysms or Abdominal Aneurysms Utilizing Fenestrated/Branched Stent-Grafts
Brief Title: Endovascular Exclusion of TAAA/AAA Utilizing Fenestrated/Branched Stent Grafts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Behzad Farivar, M. D., Principal Investigator, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G010002; IRB 4281 (Other: Cleveland Clinic IRB)
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Results first posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-04

CONDITIONS: Thoracoabdominal Aneurysm; Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Endovascular Aneurysm Repair (Experimental): Endovascular Aneurysm Repair of TAAA/AAA with Fenestrated/Branched Stent Grafts
  Interventions: Device: Endovascular Aneurysm Repair

INTERVENTIONS:
Device: Endovascular Aneurysm Repair — Endovascular exclusion of aneurysm
  Other Names: Cook Zenith

SUMMARY:
The purpose of the study is to evaluate the role of fenestrated/branched stent-grafts in the exclusion of abdominal aortic and thoracoabdominal aneurysms.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the role of fenestrated/branched stent-grafts in the exclusion of abdominal aortic and thoracoabdominal aneurysms. The evaluation shall be conducted with subjects that would be expected to have great difficulty tolerating open surgical repair and anatomies not suitable for devices currently marketed.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Not pregnant
3. Willing and able to comply with two-year follow-up period.
4. Willing and able to give informed consent prior to enrollment
5. No known allergy to stainless steel or polyester
6. No history of anaphylactic reaction to contrast material with an inability to properly prophylax the patient appropriately.
7. Life expectancy greater than two years
8. High risk candidate for open surgical repair

Exclusion Criteria:

see above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1366 (Actual)
Dates: Start 2001-02 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Behzad Farivar, M. D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang J, Brier C, Parodi FE, Kuramochi Y, Lyden SP, Eagleton MJ. Incidence and management of iliac artery aneurysms associated with endovascular treatment of juxtarenal and thoracoabdominal aortic aneurysms. J Vasc Surg. 2020 Oct;72(4):1360-1366. doi: 10.1016/j.jvs.2019.12.040. Epub 2020 Mar 12. PMID 32173192
- [Derived] Eagleton MJ, Follansbee M, Wolski K, Mastracci T, Kuramochi Y. Fenestrated and branched endovascular aneurysm repair outcomes for type II and III thoracoabdominal aortic aneurysms. J Vasc Surg. 2016 Apr;63(4):930-42. doi: 10.1016/j.jvs.2015.10.095. Epub 2016 Jan 11. PMID 26792544
- [Derived] Sylvan J, Brier C, Wolski K, Yanof J, Goel V, Kuramochi Y, Eagleton MJ. Impact of alterations in target vessel curvature on branch durability after endovascular repair of thoracoabdominal aortic aneurysms. J Vasc Surg. 2016 Mar;63(3):634-41. doi: 10.1016/j.jvs.2015.09.053. Epub 2015 Nov 29. PMID 26620715
- [Derived] Mastracci TM, Eagleton MJ, Kuramochi Y, Bathurst S, Wolski K. Twelve-year results of fenestrated endografts for juxtarenal and group IV thoracoabdominal aneurysms. J Vasc Surg. 2015 Feb;61(2):355-64. doi: 10.1016/j.jvs.2014.09.068. PMID 25619574
- [Derived] O'Callaghan A, Greenberg RK, Eagleton MJ, Bena J, Mastracci TM. Type Ia endoleaks after fenestrated and branched endografts may lead to component instability and increased aortic mortality. J Vasc Surg. 2015 Apr;61(4):908-14. doi: 10.1016/j.jvs.2014.10.085. Epub 2015 Jan 16. PMID 25600335
- [Derived] O'Callaghan A, Mastracci TM, Eagleton MJ. Staged endovascular repair of thoracoabdominal aortic aneurysms limits incidence and severity of spinal cord ischemia. J Vasc Surg. 2015 Feb;61(2):347-354.e1. doi: 10.1016/j.jvs.2014.09.011. Epub 2014 Oct 23. PMID 25449006
- [Derived] O'Callaghan A, Mastracci TM, Greenberg RK, Eagleton MJ, Bena J, Kuramochi Y. Outcomes for supra-aortic branch vessel stenting in the treatment of thoracic aortic disease. J Vasc Surg. 2014 Oct;60(4):914-20. doi: 10.1016/j.jvs.2013.12.053. Epub 2014 Jul 1. PMID 24993951
- [Derived] Eagleton MJ, Shah S, Petkosevek D, Mastracci TM, Greenberg RK. Hypogastric and subclavian artery patency affects onset and recovery of spinal cord ischemia associated with aortic endografting. J Vasc Surg. 2014 Jan;59(1):89-94. doi: 10.1016/j.jvs.2013.07.007. Epub 2013 Nov 1. PMID 24188715
- [Derived] Mohapatra A, Greenberg RK, Mastracci TM, Eagleton MJ, Thornsberry B. Radiation exposure to operating room personnel and patients during endovascular procedures. J Vasc Surg. 2013 Sep;58(3):702-9. doi: 10.1016/j.jvs.2013.02.032. Epub 2013 Jun 28. PMID 23810300
- [Derived] Brown CR, Greenberg RK, Wong S, Eagleton M, Mastracci T, Hernandez AV, Rigelsky CM, Moran R. Family history of aortic disease predicts disease patterns and progression and is a significant influence on management strategies for patients and their relatives. J Vasc Surg. 2013 Sep;58(3):573-81. doi: 10.1016/j.jvs.2013.02.239. Epub 2013 Jul 1. PMID 23809203
- [Derived] Kitagawa A, Greenberg RK, Eagleton MJ, Mastracci TM, Roselli EE. Fenestrated and branched endovascular aortic repair for chronic type B aortic dissection with thoracoabdominal aneurysms. J Vasc Surg. 2013 Sep;58(3):625-34. doi: 10.1016/j.jvs.2013.01.049. Epub 2013 Jun 22. PMID 23800455
- [Derived] Kitagawa A, Greenberg RK, Eagleton MJ, Mastracci TM. Zenith p-branch standard fenestrated endovascular graft for juxtarenal abdominal aortic aneurysms. J Vasc Surg. 2013 Aug;58(2):291-300. doi: 10.1016/j.jvs.2012.12.087. Epub 2013 Apr 20. PMID 23611709
- [Derived] Mastracci TM, Greenberg RK, Eagleton MJ, Hernandez AV. Durability of branches in branched and fenestrated endografts. J Vasc Surg. 2013 Apr;57(4):926-33; discussion 933. doi: 10.1016/j.jvs.2012.09.071. Epub 2013 Feb 20. PMID 23433817

RESULTS

PARTICIPANT FLOW:
Groups:
- Endovascular Aneurysm Repair: Treatment Arm: Subjects with abdominal/thoracoabdominal aneurysm undergoing endovascular aneurysm repair
Period: Overall Study
Arm/Group | Endovascular Aneurysm Repair
Started | 1366
Completed | 1366
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Endovascular Aneurysm Repair
Number analyzed (Participants) | 1366
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 141
  >=65 years | 1225
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 315
  Male | 1051
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 1366
Presence of abdominal or thoracoabdominal aneurysm [Count of Participants; unit: Participants] | 1366

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Aneurysm Rupture
Description: Absence of blood extravasation outside of aneurysm sac demonstrated by CT scan
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Endovascular Aneurysm Repair
Number analyzed (Participants) | 1366
Participants | 22

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Endovascular Aneurysm Repair
All-Cause Mortality (participants affected / at risk) | 775/1366
Serious Adverse Events (participants affected / at risk) | 22/1366
Other Adverse Events (participants affected / at risk) | 68/1366
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Endovascular Aneurysm Repair (N=1366)
Aneurysm Rupture (Vascular disorders) | 22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Endovascular Aneurysm Repair (N=1366)
Aneurysm size increase (Vascular disorders) | 68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT00583050/Prot_000.pdf
  • Statistical Analysis Plan (2006-03-09): https://cdn.clinicaltrials.gov/large-docs/50/NCT00583050/SAP_001.pdf
  • Informed Consent Form (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT00583050/ICF_002.pdf